CLINICAL TRIAL: NCT06927583
Title: Effect of Sensory Integration in Speech Therapy for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0659
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory integration therapy (Experimental): Experimental group was given sensory integration therapy .total number of 5 sessions give t o each participant that comprised of 30 minutes.
  Interventions: Other: sensory integration therapy
- Traditional Speech therapy (Active Comparator): Control group was given traditional speech therapy .total number of 5 sessions give t o each participant that comprised of 30 minutes.
  Interventions: Other: Traditional Speech therapy

INTERVENTIONS:
Other: sensory integration therapy — sensory integration therapy include 2 categories that comprised of 9 strategies.
  Other Names: Traditional speech therapy
  Arms: Sensory integration therapy
Other: Traditional Speech therapy — Control group was given traditional speech therapy .total number of 5 sessions give t o each participant that comprised of 30 minutes.
  Arms: Traditional Speech therapy

SUMMARY:
Autism spectrum disorder (ASD) is considered one of the commonest developmental disabilities, characterized mainly by impairments in social performance and communicative skills, repetitive stereotypical behaviors, and restriction in interests and activities, with a combination of sensory, cognitive, behavioral, and communication features which persist throughout life. Caminha & Lampreia specified that there is a significantly high prevalence of sensory processing dysfunctions in ASD. Sensory processing means how the central and peripheral nervous systems deal with the incoming sensory input from different sensory organs; visual, auditory, smell, taste, tactile, proprioception, and vestibular information. Sensory processing dysfunction is the neurological dysfunction affecting the adequate reception, modulation, integration, discrimination, or organization of sensory stimuli, and the behavioral responses to the sensory input. Sensory integration therapy (SIT) is a frequent type of therapy that aims to improve a child's ability to perceive and integrate sensory input in order to explore more ordered and appropriate actions. SIT improves motor skills, social relationships, attention, behavior control, language and pre-linguistic communicative abilities, reading comprehension, participation in play activities, and personal identification. Therefore, the need for further explicit assessment of sensory integration intervention among ASD children has been increased to identify its gains in social and verbal interactions. This study aimed to estimate the impact of sensory integration therapy on language development in autism spectrum disorder children.46 ASD children will enroll in this study, their ages ranged from 3-10 years, males and females, divided into two groups (group I received speech therapy sessions together with sensory integration therapy sessions, group II received speech therapy sessions only) went through two stages of evaluation before and after receiving their sessions with one year apart. All children were subjected to Childhood Autism Rating Scale (CARS), sensory profile assessment by Short Sensory profile (SSP) and Assessment of Basic Language and Learning Skills- Revised (The ABLLS-R).Data will be taken from Clinics and Schools having children with autism

ELIGIBILITY:
Inclusion Criteria:

* Pre diagnosed autistic children
* Both male and female
* Age range:3 years to 10 years
* Moderately severe

Exclusion Criteria:

- Autism with any comorbid will be excluded ( hearing impaired, Any syndrome)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Basic Language and Learning Skills- Revised (ABLLS-R) | baseline and 6 weeks
  The ABLLS-R scoring system evaluates a child's skills across 25 developmental areas. Each task within a skill area is broken into steps, scored on a 0-2 scale: 0 for no skill, 1 for emerging or assisted performance, and 2 for independent mastery. The scores for all steps in a task are totaled to give a task score, which contributes to the overall skill area score. A visual tracking grid is used to record and color-code performance, helping identify strengths, areas for improvement, and track progress over time. This scoring guides individualized goal setting and intervention planning.

CONTACTS AND LOCATIONS:
Overall Officials: Hina Omer, Ms(SLP), Principal Investigator — Riphah International University
Locations (1):
- Hayyati Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barros VdM, Folha DRdSC, Pinheiro RC, Della Barba PCdSJCBdTO. Sensory processing and engagement: a systematic review. 2023;31:e3521.
- [Background] Randell E, Wright M, Milosevic S, Gillespie D, Brookes-Howell L, Busse-Morris M, Hastings R, Maboshe W, Williams-Thomas R, Mills L, Romeo R, Yaziji N, McKigney AM, Ahuja A, Warren G, Glarou E, Delport S, McNamara R. Sensory integration therapy for children with autism and sensory processing difficulties: the SenITA RCT. Health Technol Assess. 2022 Jun;26(29):1-140. doi: 10.3310/TQGE0020. PMID 35766242